CLINICAL TRIAL: NCT06446973
Title: Evaluation Of Pain, Balance, Functional Performance and Quality of Life in Patients With Meniscus Lesions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Aydın University (Other)
Responsible Party: Principal Investigator, Barış CELBEK, Lecturer, Istanbul Aydın University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Istanbula
Record Dates: First submitted 2024-06-01; First posted 2024-06-06 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-06

CONDITIONS: Meniscus Tear; Quality of Life
Keywords: Peniscus tear; Pain; Quality of Life; Balance; Muscle Strenght
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): 35 healthy individuals
- Meniscus tear group (Active Comparator): 35 patients diagnosed with meniscus tear
  Interventions: Other: 35 patients with meniscus tear

INTERVENTIONS:
Other: 35 patients with meniscus tear — Have meniscus pathologies in one or both knees confirmed by MRI.
  Arms: Meniscus tear group

SUMMARY:
Meniscal tears are common knee injuries, affecting a wide demographic from young athletes to the elderly population, often resulting from traumatic sports-related incidents or degenerative processes associated with aging. The impact of meniscal injuries extends beyond the immediate physical damage, influencing pain perception, balance, functional performance, and ultimately, the quality of life. Despite advancements in diagnostic and therapeutic strategies, the comprehensive effects of meniscal tears on these domains remain inadequately explored, particularly regarding their correlation with objective measures of pain, balance, muscle strength and quality of life.

The meniscus plays a crucial role in knee joint stability, load distribution, and shock absorption. Damage to this fibrocartilaginous structure can significantly impair knee function, leading to altered biomechanics, decreased joint stability, and increased risk of osteoarthritis. Previous research has predominantly focused on the surgical and non-surgical management of meniscal tears, with less attention to the broader implications on patients' daily lives, particularly in terms of postural stability, risk of falls, and overall physical well-being.

This study aims to bridge this knowledge gap by quantitatively assessing the risk of meniscal tears on pain levels, balance, functional performance, and quality of life. By comparing objective measurements between individuals with meniscal tears and healthy controls, the investigators seek to elucidate the multifaceted impact of these injuries. Understanding these relationships is crucial for developing targeted rehabilitation strategies that address not only the mechanical aspects of the injury but also the associated functional and quality of life concerns.

Our hypothesis was that individuals with meniscal lesions have worse pain, functional performance and quality of life compared to those without such injuries and also pain directly influences balance, functional performance, and quality of life in patients with meniscal injuries.

DETAILED DESCRIPTION:
This study included a total of 70 participants, divided into two groups: 35 patients diagnosed with meniscus tear and 35 healthy individuals. The investigators determined this sample size using the G-Power software to ensure a 95% power level and an effect size of 0.8, following the methodology recommended by Faul et al.

The criteria for inclusion in the meniscopathy group;

* Volunteering to participate in the research,
* To be between ages of 18-60,
* Not having systemic or neurological issues interfering with assessment completion,
* Have meniscus pathologies in one or both knees confirmed by MRI.

The criteria for inclusion in the control group;

* To be between ages of 18-60,
* Not have any orthopedic, neurological, or systemic conditions, Volunteer to participate in the study. Exlusion criteria from the study;
* Having had additional knee surgery or fractures in the affected lower extremity within the last year
* Having had autoimmune or inflammatory diseases,
* Having had involved in a physiotherapy program for the knee in the past six months.

Physical Properties and Sociodemographic Assessment Age, sex, height, body weight, dominant lower extremity, occupation was recorded. In addition, the affected side, the duration of complaints, and insights into the participants' activity levels and habits were noted.

Pain Severity and Range of Motion Assessment Pain intensity was quantified using the Visual Analog Scale (VAS), during various states such as activity, rest, and nighttime. Joint Range of Motion (ROM) was evaluated with a goniometer, adhering to established protocols for knee flexion and extension, to increase reliability in our measurements.

Muscle Strength Assessment Hamstring muscle group and Quadriceps Femoris muscle were evaluated. The knee flexion and extension muscle strengths of the subjects were given a value between 0 and 5 according to the resistance applied to the muscle in standard positions

Balance Assessment Berg Balance Scale (BBS) was utilized to determine fall risk and postural control. This test has a 14-item test that is used to assess the self-perceived balance among individuals. The total score ranges between 0 and 56, with higher scores indicating a better balance. The validity and reliability study of the Turkish version of BBS has been studied

Physical Performance Assessment Physical performance was further assessed via the Timed Up and Go Test (TUG) and the Five Times Sit to Stand Test (5TSTS) , both of which measure balance, walking speed, and functional mobility by timing participants in task-specific movements. For the TUG test, a point 3 m away from the participant's chair was marked and the participant was asked to get up from the chair, walk 3 m, return and sit back down and the completion time of the test was measured with a stopwatch. Participants were instructed to wear comfortable shoes. 5TSTS ; In this test, the patient sat with arms crossed over the chest and back against the chair. Upon the command "Start," the patient was asked to quickly stand up and sit down from a standard chair five times. The elapsed time was measured with a stopwatch and recorded in seconds.

Quality of Life Assessment The quality of life for those with meniscus pathology was evaluated using the Western Ontario Meniscal Evaluation Tool (WOMET), a Turkish-validated questionnaire that segments 16 questions into physical symptoms, lifestyle/work, and emotional impact, providing a comprehensive view of the participants' well-being.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the research,
* To be between ages of 18-60,
* Not having systemic or neurological issues interfering with assessment completion,
* Have meniscus pathologies in one or both knees confirmed by MRI.

The criteria for inclusion in the control group;

* To be between ages of 18-60,
* Not have any orthopedic, neurological, or systemic conditions,
* Volunteer to participate in the study.

Exclusion Criteria:

* - Having had additional knee surgery or fractures in the affected lower extremity within the last year
* Having had autoimmune or inflammatory diseases,
* Having had involved in a physiotherapy program for the knee in the past six months.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Pain Severity and Range of Motion Assessment | through study completion, an average of 1 year
  Pain intensity was quantified using the Visual Analog Scale (VAS), during various states such as activity, rest, and nighttime. Joint Range of Motion (ROM) was evaluated with a goniometer, adhering to established protocols for knee flexion and extension, to increase reliability in our measurements.There are numbers from 0 to 10. 0 is classified as no pain and 10 as very severe.
Muscle Strength Assessment | through study completion, an average of 1 year
  Hamstring muscle group and Quadriceps Femoris muscle were evaluated.The knee flexion and extension muscle strengths of the subjects were given a value between 0 and 5 according to the resistance applied to the muscle in standard positions
Balance Assessment | through study completion, an average of 1 year
  Berg Balance Scale (BBS) was utilized to determine fall risk and postural control.This test has a 14-item test that is used to assess the self-perceived balance among individuals. The total score ranges between 0 and 56, with higher scores indicating a better balance.
Physical Performance Assessment- TUG | through study completion, an average of 1 year
  Timed Up and Go Test (TUG ). For the TUG test, a point 3 m away from the participant's chair was marked and the participant was asked to get up from the chair, walk 3 m, return and sit back down and the completion time of the test was measured with a stopwatch
Physical Performance Assessment- 5TSTS | through study completion, an average of 1 year
  Participants were instructed to wear comfortable shoes. 5TSTS ; In this test, the patient sat with arms crossed over the chest and back against the chair. Upon the command "Start," the patient was asked to quickly stand up and sit down from a standard chair five times. The elapsed time was measured with a stopwatch and recorded in seconds.
Quality of Life Assessment | through study completion, an average of 1 year
  The quality of life for those with meniscus pathology was evaluated using the Western Ontario Meniscal Evaluation Tool (WOMET).a Turkish-validated questionnaire that segments 16 questions into physical symptoms, lifestyle/work, and emotional impact, providing a comprehensive view of the participants' well-being

CONTACTS AND LOCATIONS:
Locations (1):
- Barış CELBEK, Istanbul, Turkey (Türkiye)